CLINICAL TRIAL: NCT04367220
Title: Cardiovascular Imaging Registry of Canada
Acronym: CIROC
Status: Recruiting | Type: Observational
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Principal Investigator, James White, MD, FRCP(C) Director - Stephenson Cardiac Imaging Centre, University of Calgary
Other Study IDs: REB13-0902
Record Dates: First submitted 2020-04-26; First posted 2020-04-29 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with known or suspected cardiovascular disease: All patients with known or suspected cardiovascular disease are studied with a-priori stratification of specific disease-based cohorts.
  Interventions: Diagnostic Test: Diagnostic testing performed as per routine care

INTERVENTIONS:
Diagnostic Test: Diagnostic testing performed as per routine care

SUMMARY:
A multi-site, multi-modality prospective observational clinical outcomes study focussed on the development of phenotype-dirven risk prediction modelling in patients with known or suspected cardiovascular disease.

DETAILED DESCRIPTION:
The Cardiovascular Imaging Registry of Canada (CIROC) was conceived to provide a common standardized architecture for the collection of clinically reported imaging biomarkers, demographic information, resource utilization and clinical outcomes among patients referred to non-invasive cardiac imaging. The Registry was designed to assess the feasibility of implementing personalized care strategies through automated high quality data collection and patient engagement.

The CIROC Registry was launched with inaugural focus on Cardiac MRI base phenotyping, however has evolved to encompass cardiac CTA and echocardiography. Clinically referred patients are engaged by automated, tablet-based tools to collect informed consent and deploy standardized patient health assessments. Standardized reporting of disease features are captured using bespoke reporting tools. All patients are prospectively followed for a period of 10-years using linkage to administrative health data, inclusive of ICD-coded events, laboratory test results, ECG and vital statistics.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for hospital-based cardiac imaging services

Exclusion Criteria:

* Failure or provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred for hospital based cardiac imaging services are considered eligible and are routinely approached using automated patient engagement tools and consent management services.
Sampling Method: Non-Probability Sample
Enrollment: 45000 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular outcomes (MACE) | 2024
  Composite of all-cause death, heart failure admission, myocardial infarction, heart transplantation or LVAD, Stroke or TIA
Malignant arrhythmic events | 2024
  Composite of sudden cardiac death or appropriate ICD shock
Heart failure events | 2024
  Composite of heart failure admission, death or need for transplantation / LVAD
Atrial arrhythmic events | 2024
  Occurrence of atrial fibrillation / atrial flutter (documented by 12-lead ECG or Holter monitor)
All-cause mortality | 2024
  Death based on Vital Statistics Alberta and In-hospital coded death

CONTACTS AND LOCATIONS:
Overall Officials: James White, Principal Investigator — Director of Stephenson Cardiac Imaging Centre
Locations (4):
- Canada (4):
  - Foothills Medical Centre, Calgary, Alberta
  - South Health Campus, Calgary, Alberta
  - Peter Lougheed Hospital, Calgary, Alberta
  - Rockyview Hospital, Calgary, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Purmah Y, Lei LY, Dykstra S, Mikami Y, Cornhill A, Satriano A, Flewitt J, Rivest S, Sandonato R, Seib M, Lydell CP, Howarth AG, Heydari B, Merchant N, Bristow M, Fine N, Gaztanaga J, White JA. Right Ventricular Ejection Fraction for the Prediction of Major Adverse Cardiovascular and Heart Failure-Related Events: A Cardiac MRI Based Study of 7131 Patients With Known or Suspected Cardiovascular Disease. Circ Cardiovasc Imaging. 2021 Mar;14(3):e011337. doi: 10.1161/CIRCIMAGING.120.011337. Epub 2021 Mar 16. PMID 33722059